CLINICAL TRIAL: NCT01812031
Title: Benefits Study of a Respiratory Gating Protocol for Positron Emission Tomography: Application on the Lungs
Brief Title: Benefits Study of Respiratory-gated PET Acquisition in Lung Disease
Acronym: PneumoTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: AOL09-PR-MEYER; 2009-A00491-56 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer; Chronic Obstructive Pulmonary Disease
Keywords: PET/CT; 18F-fluoro-2-deoxyglucose; lung neoplasms; respiratory motion
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Pulmonary Disease, Chronic Obstructive | interventions — X-Rays

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lung nodules (Experimental): "Medical imaging" intervention applied on patients included in the trial
  Interventions: Other: medical imaging

INTERVENTIONS:
Other: medical imaging — After fasting for at least 6 hours, normal glucose blood level was checked and each patient received an intravenous injection of 18F-FDG (5MBq/kg). After a 60-minute uptake phase in a quiet environment, patients underwent the PET/CT examination.
  Whole-body PET/CT (Ungated session) The Ungated acquisition consisted in a whole-body, free-breathing CT followed by standard multistep PET, used as routine clinical practice in the department.
  Respiratory-gated PET/CT (CT-based session) The CT-based method consisted in an additional single-step, 10-minute List Mode respiratory gated PET acquisition followed by an end-expiration breath-hold CT added to the end of the clinical protocol, with continuous respiratory signal recording during these examinations.
  Other Names: Biograph; Siemens medical solutions; Anzai medical

SUMMARY:
Fluorodeoxyglucose (FDG) positron emission tomography (PET) is now widely used for cancer imaging purpose, notably for preoperative work-up. It aims at visualizing organs metabolism. In case of cancer, metabolism is, classically, increased and some hot spots are visible on PET images. Because of respiratory motion some lung tumours (especially the smallest ones) can be falsely interpreted by the clinician.

The investigators developed a respiratory-gated PET method in order to reduce the motion issue. The investigators designed a study to investigate its effect on lung cancer (primary or metastasis) to check if it improves the sensitivity/specificity of PET imaging of the lungs.

To that aim, patients presenting a lung nodule on a CT examination can be proposed to participate this study. After the standard PET acquisition (acquired in free-breathing), an additional 10 minutes respiratory-gated PET acquisition is performed without additional injection. After that, a breath-hold (~10s) CT is performed.

ELIGIBILITY:
Inclusion Criteria:

* patient has one or more lung lesion(s) less than 35 mm visible on a CT image
* age : over 18 years
* patients gave their written informed consent

Exclusion Criteria:

* pregnancy
* patient has at least one lesion more than 35 mm in its great axis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-08; Primary Completion 2013-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Lesion SUVmax | Day 1
  For each CT nodule, observer has to report the corresponding (maximum Standardized Uptake Value)SUVmax on ungated and CT-based images (even if there is no obvious uptake)

SECONDARY OUTCOMES:
Lung function test | Day 0
  Patients undergo lung function test including measures of:
  * total lung capacity
  * residual volume
  * forced expiratory volume
  * forced vital capacity

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Etienne MEYER, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, Picardie, France

REFERENCES:
- [Result] Daouk J, Leloire M, Fin L, Bailly P, Morvan J, El Esper I, Saidi L, Moullart V, Francois G, Jounieaux V, Meyer ME. Respiratory-gated 18F-FDG PET imaging in lung cancer: effects on sensitivity and specificity. Acta Radiol. 2011 Jul 1;52(6):651-7. doi: 10.1258/ar.2011.110018. Epub 2011 Apr 21. PMID 21511870
- [Result] Daouk J, Bailly P, Kamimura M, Sacksick D, Jounieaux V, Meyer ME. Positron emission tomography-based evidence of low-amplitude respiratory motion in patients with chronic obstructive pulmonary disease. Ann Nucl Med. 2015 May;29(4):319-24. doi: 10.1007/s12149-014-0945-3. Epub 2015 Jan 8. PMID 25567204
- [Result] Fin L, Daouk J, Morvan J, Bailly P, El Esper I, Saidi L, Meyer ME. Initial clinical results for breath-hold CT-based processing of respiratory-gated PET acquisitions. Eur J Nucl Med Mol Imaging. 2008 Nov;35(11):1971-80. doi: 10.1007/s00259-008-0858-2. Epub 2008 Jun 26. PMID 18581114